CLINICAL TRIAL: NCT04795700
Title: Effects of Mindfulness Self-Compassion Intervention on the Dyadic Mental Health of Lung Cancer Patients and Their Caregivers: a Randomized Controlled Trial
Brief Title: Effects of MSC Intervention on the Dyadic Mental Health of Lung Cancer Patients and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Juan LI, Principal investigator, Central South University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MSC
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Depression, Anxiety
Keywords: lung cancer patients; caregivers; mindfulness; self-compassion; resilience; intimacy
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Patients in the intervention group had access to conventional care, in addition to receiving the follow-up MSC intervention sessions. The intervention was provided by trained nurses, including one researcher and one MSC therapist. The researcher was regarded as primary leader of the intervention sessions. The leader informed patients of the schedule for each session using the educational manual 'Caring for ourselves, we are together' (developed by psychologists, nursing managers, experienced oncology nurses, and researchers).
  No interventions were performed for the control group participants during the study. However, these patients received conventional care in the oncology departments according to the two hospitals' similar nursing guidelines.
Who Masked: Participant, Outcomes Assessor
Masking Description: Potential eligible participants were identified by researchers according to medical records at the oncology departments in each hospital. They were recruited with informed consent, and researchers explained the study purposes, procedures, benefits, and risks involved orally. The participants were then randomly allocated to the intervention or the control group according to a computer-generated block randomization list. The generated random numbers were put into consecutively numbered and opaque sealed envelopes. When enrolling and randomising a new participant, the enrolling investigators opened the sealed envelope after participant's name was written on next available envelopes. A sequentially numbered and opaque , sealed envelope system was used by a non-investigator. Additionally, all data collection was conducted by another research assistant who was blind to the study design and allocation of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): Patients in the intervention group receiving the 8 weeks MSC intervention sessions.
  Interventions: Behavioral: MSC intervention
- The control group (No Intervention): No interventions except conventional care were performed for the control group.

INTERVENTIONS:
Behavioral: MSC intervention — Patients in the intervention group had access to conventional care, in addition to receiving the 8 weeks MSC intervention sessions. The intervention was provided by trained nurses, including one researcher and one MSC therapist. The intervention is mainly out-of-hospital intervention, supplemented by short-term in-hospital intervention. Among them, the first and second weeks of the intervention project in the hospital phase focus on guiding the research subjects to understand the content of mindful self-compassion and emotions, and carry out basic mindful self-compassion training; the content of the 3-8th week of the intervention program outside the hospital, Focus on the maintenance of mindful self-compassion training and the promotion of mindful life. Each face-to-face group contact lasted about 1 hour, depending on the complexity of the patients' problems.
  Arms: The intervention group

SUMMARY:
The incidence and mortality of lung cancer ranks first among cancers in the world, and the five-year survival rate of lung cancer patients is only 15% to 30%. Lung cancer patients bear a great psychological pressure, prone to anger, isolation, anxiety, depression, self-esteem and other psychological problems. The incidence of psychological disorders in lung cancer patients was 24.2 to 73.4%. A diagnosis of cancer not only causes physical and mental pain to the patient, but also has a huge impact on the family and their caregivers. As patients'primary coping resources, caregivers have to bear both physical and mental pressures. Therefore, it is worth to attention the mental health of lung cancer patients and their caregivers.

With the further deepening of self-concept research and the integration of Buddhist thought and psychology, the new concept of 'self-compassion' was proposed and developed. Self-compassion means that individuals treat themselves like their friends, with a friendly and tolerant attitude; maintains an objective and rational attitude towards the individual's own situation at all times; thinks that pain is a common experience shared by others, and everyone should be understood and sympathized. At the same time, self-compassion not only includes acceptance and affirmation of oneself, but also connects oneself with others, advocating that one should sympathize with oneself as sympathizing with others, providing the possibility of emotional connection between patients and their caregivers. Therefore, the study of mindfulness and self-compassion is expected to provide a reference for improving the dyadic mental health of lung cancer patient-caregiver dyads in China.

Mindfulness Self-Compassion (MSC) is a positive psychology intervention method that covers the concept of self-compassion developed by Neff and Germer on the basis of Mindfulness-based Stress Reduction. MSC is a 2.5-hour weekly, 8-week standardized training course. Some studies have shown that MSC can promote the emotional health of cancer patients and buffer their mental symptoms.

To sum up, the current mindfulness self-compassion training program has been applied to some cancer patients, and shows that the intervention has a positive effect, while the research in China has only been initially applied in the student population, and has not been applied in the field of cancer. Therefore, for lung cancer patient-caregiver dyad, the researchers can learn from the experience of mindfulness self-compassion training and develop a dyadic mental health intervention program based on Chinese condition. The current study aims to verify the effect of the dyadic mindfulness self-compassion intervention program for lung cancer patients and their caregivers, and explore its mechanism.

DETAILED DESCRIPTION:
The study was a single blind, follow-up, randomized, controlled trial. Researchers recruited subjects from two general tertiary hospitals in Changsha, Hunan province, China. And the whole trail was on the basis of the CONSORT statements. The two hospitals provided similar conventional care for lung cancer patients. Study procedures were approved by the institutional review boards of all participating centers before data collection began. All patients were screened by researchers for eligibility and then enrolled in the study if eligible and if the provided consent.

Potential eligible participants were identified by researchers according to medical records at the colorectal surgery unit in each hospital. The participants were recruited with informed consent, and researchers explained the study purposes, procedures, benefits, and risks involved orally. The participants were then randomly allocated to the intervention or the control group according to a computer-generated block randomization list. A sequentially numbered and opaque , sealed envelope system was used by a non-investigator. The generated random numbers were put into consecutively numbered and opaque sealed envelopes. When enrolling and randomising a new participant, the enrolling investigators opened the sealed envelope after participant's name was written on next available envelopes; the enrolling investigators were blinded to the trial design and study hypotheses.

The researcher will recruit 74 lung cancer patient-caregiver dyads and randomly divide them into 2 groups: the control group, the dyadic intervention group. Among them, patients in the control group and caregivers received routine psychological care programs; patients in the intervention group had access to conventional care, in addition to receiving the 8-week dyadic MSC intervention sessions. The intervention was provided by trained nurses, including one researcher and one MSC therapist. The researcher was regarded as primary leader of the intervention sessions. The leader informed patients of the schedule for each session using the educational manual'Caring for ourselves, we are together' (developed by psychologists, nursing managers, experienced MSC therapist, oncology Nurse, and researchers).

The MSC techniques include body scanning, breathing meditation, sitting meditation, walking meditation, loving-kindness practice, and self-compassion writing expression. Intensive training once a week, 1 hour each time, encourage students to use 15-20 minutes a day to learn these skills, the total training time per week is 2.5 hours. The intervention is mainly out-of-hospital intervention, supplemented by short-term in-hospital intervention (1-2 weeks, adjusted according to the patient's hospital stay). The in-hospital stage focuses on guiding the research subjects to understand the content of mindful self-compassion and emotions, and conduct basic mindful self-compassion training; the outside of the hospital focuses on the maintenance of mindful self-compassion training and the promotion of mindful life.

Data were collected by a research assistant who was blind to the study design and allocation of participants. At baseline, before randomization, sociodemographic and clinical characteristics were collected from medical records and personal interviews. The two groups of participants completed surveys after each follow-up via face to face interviews at baseline (T0) and immediately after intervention (T1). The next two evaluations were performed at 1-month (T2) and 3-months (T3) after intervention via telephone contact.

ELIGIBILITY:
For lung cancer patients

Inclusion Criteria:

* Diagnosed with lung cancer by pathological biopsy or cytology;
* The disease condition is relatively stable;
* Must be conscious, with normal communication ability;
* Must be volunteered to join the study.

Exclusion Criteria:

* Share a hospital room with a current study participant;
* With other types of cancer;
* Alcoholics and/or drug addicts;
* Disabilities and cannot take care of themselves.

For caregivers

Inclusion Criteria:

* A primary caregiver designated by a lung cancer patient who has been included in this study, with a cumulative care time of more than 72 hours;
* One of the family members of a hospitalized lung cancer patient, such as their spouse, children, parents or other relatives
* must be conscious, with normal communication ability;
* must be volunteered to join the study.

Exclusion Criteria:

* Have an employment relationship with the patient, such as nurses and nanny；
* Alcoholics and/or drug addicts;
* Disabilities and cannot take care of themselves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Depression of lung cancer patients and their caregivers | 3-months (T3) after intervention
  Patient Health Questionnaire 2-item Depression Screen (PHQ-2) is used to initially screen the high-risk groups of depression. The score of each item ranges from "0 means no at all" to "3 points means almost every day". The total score is equal to the sum of the items is 6 points, and 3 points or more can be considered as depressed. . PHQ-2 has good reliability and validity in the screening of depression in patients with cardiovascular diseases. Cronbach's α coefficient is 0.809, and the test-retest reliability coefficient is 0.882.
Anxiety of lung cancer patients and their caregivers | 3-months (T3) after intervention
  Generalized Anxiety Disorder-7 (GAD-7) is used to screen for Generalized Anxiety. There are 7 items in total. It is scored from 0 (never) to 3 (almost every day). , The higher the score, the more serious the anxiety. According to Spitzer's assessment of GAD-7 scale, 5 is divided into the cut-off value of symptom-positive samples.

SECONDARY OUTCOMES:
Self-compassion of lung cancer patients and their caregivers | 3-months (T3) after intervention
  The Self-compassion Scale has good adaptability in both healthy people and patients with chronic diseases. The scale contains 6 subscales of self-tolerance, self-criticism, universal humanity, loneliness, mindfulness and over-identification, with a total of 26 items. Each item uses a Likert 5-level score, ranging from "never" to "always". The score is 1 to 5, and the total score is 26 to 130. The three dimensions of self-criticism, loneliness, and over-identification use the reverse scoring method. The Cronbach coefficient of the scale is 0.84, and the test-retest reliability is 0.89.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangtan Central Hospital, Xiangtan, Hunan, China

IPD SHARING:
Plan to Share IPD: No
The process of data collection cost a lot of human and material resources, some of the data was privacy information of participants, and so on. Considering this, it is improper to share these data.

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Mitsudomi T, Takahashi T. [Genetic abnormalities in lung cancer and their prognostic implications]. Gan To Kagaku Ryoho. 1996 Jul;23(8):990-6. Japanese. PMID 8687234
- [Background] Hamer M, Chida Y, Molloy GJ. Psychological distress and cancer mortality. J Psychosom Res. 2009 Mar;66(3):255-8. doi: 10.1016/j.jpsychores.2008.11.002. Epub 2009 Jan 16. PMID 19232239
- [Background] Qureshi F, Shafi A, Ali S, Siddiqui N. Clinical predictors of anticipatory emesis in patients treated with chemotherapy at a tertiary care cancer hospital. Pak J Med Sci. 2016 Mar-Apr;32(2):337-40. doi: 10.12669/pjms.322.9493. PMID 27182235
- [Background] Chad-Friedman E, Coleman S, Traeger LN, Pirl WF, Goldman R, Atlas SJ, Park ER. Psychological distress associated with cancer screening: A systematic review. Cancer. 2017 Oct 15;123(20):3882-3894. doi: 10.1002/cncr.30904. Epub 2017 Aug 22. PMID 28833054
- [Background] Thomas BC, NandaMohan V, Nair MK, Pandey M. Gender, age and surgery as a treatment modality leads to higher distress in patients with cancer. Support Care Cancer. 2010 Feb;19(2):239-50. doi: 10.1007/s00520-009-0810-4. Epub 2010 Feb 23. PMID 20174987
- [Background] Lee YH, Liao YC, Shun SC, Lin KC, Liao WY, Chang PH, Jhang SY, Yu CJ, Yang PC, Hsieh PY, Lai YH. Trajectories of caregiver burden and related factors in family caregivers of patients with lung cancer. Psychooncology. 2018 Jun;27(6):1493-1500. doi: 10.1002/pon.4678. Epub 2018 Mar 30. PMID 29476636
- [Background] Talbot F, Theriault J, French DJ. Self-Compassion: Evaluation of a Psychoeducational Website. Behav Cogn Psychother. 2017 Mar;45(2):198-203. doi: 10.1017/S1352465816000230. Epub 2016 Jun 15. PMID 27302088
- [Background] Sung MR, Patel MV, Djalalov S, Le LW, Shepherd FA, Burkes RL, Feld R, Lin S, Tudor R, Leighl NB. Evolution of Symptom Burden of Advanced Lung Cancer Over a Decade. Clin Lung Cancer. 2017 May;18(3):274-280.e6. doi: 10.1016/j.cllc.2016.12.010. Epub 2017 Jan 5. PMID 28185791
- [Background] Lin S, Chen Y, Yang L, Zhou J. Pain, fatigue, disturbed sleep and distress comprised a symptom cluster that related to quality of life and functional status of lung cancer surgery patients. J Clin Nurs. 2013 May;22(9-10):1281-90. doi: 10.1111/jocn.12228. PMID 23574291
- [Background] Schellekens MPJ, Karremans JC, van der Drift MA, Molema J, van den Hurk DGM, Prins JB, Speckens AEM. Are Mindfulness and Self-Compassion Related to Psychological Distress and Communication in Couples Facing Lung Cancer? A Dyadic Approach. Mindfulness (N Y). 2017;8(2):325-336. doi: 10.1007/s12671-016-0602-0. Epub 2016 Sep 6. PMID 28360948
- [Background] Toplu-Demirtas E, Kemer G, Pope AL, Moe JL. Self-compassion matters: The relationships between perceived social support, self-compassion, and subjective well-being among LGB individuals in Turkey. J Couns Psychol. 2018 Apr;65(3):372-382. doi: 10.1037/cou0000261. PMID 29672086
- [Background] Manne SL, Siegel S, Kashy D, Heckman CJ. Cancer-specific Relationship Awareness, Relationship Communication, and Intimacy Among Couples Coping with Early Stage Breast Cancer. J Soc Pers Relat. 2014 May;31(3):314-334. doi: 10.1177/0265407513494950. PMID 25242854
- [Background] Rusu PP, Hilpert P, Beach SR, Turliuc MN, Bodenmann G. Dyadic coping mediates the association of sanctification with marital satisfaction and well-being. J Fam Psychol. 2015 Dec;29(6):843-9. doi: 10.1037/fam0000108. Epub 2015 Jul 6. PMID 26147936
- [Derived] Li J, Zhou T, Li C, Zou J, Zhang J, Yuan B, Zhang J. Development of a dyadic mindfulness self-compassion intervention for patients with lung cancer and their family caregivers: A multi-method study. Asia Pac J Oncol Nurs. 2024 Nov 15;12:100622. doi: 10.1016/j.apjon.2024.100622. eCollection 2025 Dec. PMID 39712511